CLINICAL TRIAL: NCT03376789
Title: A Randomized, Multi-center, Double-Blind, Parallel-Group Clinical Study Comparing the Efficacy and Safety of MYL-1501D Produced by Two Manufacturing Processes in Type 1 Diabetes Mellitus Patients
Brief Title: Mylan Insulin Glargine Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Mylan GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MYL-1501D-3004
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Results first posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MYL-1501D (Process V Product) (Active Comparator): MYL-1501D (Process V Product)
  Interventions: Drug: MYL-1501D product using manufacture process V
- MYL-1501D (Process VI Product) (Active Comparator): MYL-1501D (Process VI Product)
  Interventions: Drug: MYL-1501D product using manufacture process VI

INTERVENTIONS:
Drug: MYL-1501D product using manufacture process V — MYL-1501D product using manufacture process V
  Arms: MYL-1501D (Process V Product)
Drug: MYL-1501D product using manufacture process VI — MYL-1501D product using manufacture process VI
  Arms: MYL-1501D (Process VI Product)

SUMMARY:
The aim of this study is to demonstrate similar efficacy and safety between MYL-1501D products produced from two manufacturing processes (Process V and Process VI) in combination with insulin lispro in patients with type 1 diabetes mellitus (T1DM).

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, parallel-group Phase 3 study in subjects with type 1 diabetes mellitus (T1DM) comparing the efficacy, immunogenicity, and safety of MYL-1501D products from 2 manufacturing processes (Process V and Process VI). After a 2-week screening period, all subjects will be titrated on Lantus® during a 4-week run-in period and shifted from their current mealtime insulin to insulin lispro (Humalog®). Subjects will then be randomized (stratified by time of administration of glargine [morning and evening]) to 1 of 2 groups:

* MYL-1501D product from Process V
* MYL-1501D product from Process VI Treatment with MYL-1501D is for 18 weeks. A follow-up visit is scheduled 2 weeks after last dose of MYL 1501D.

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent needs to be provided by subjects or their legal representatives before starting any protocol-specific procedures.
2. Male and female subjects between the ages of 18 to 65 years, both ages inclusive.
3. Subjects with an established diagnosis of T1DM per ADA 2017 criteria who also fulfil the following criteria:

   1. Initiation of insulin treatment within 6 months of T1DM diagnosis
   2. Treatment with basal-bolus insulin therapy for at least 1 year before screening
   3. Fasting plasma C-peptide <0.3 nmol/L at screening
   4. Subject has been on once daily Lantus® at stable dose (±15% variation in dose) for at least 3 months at screening
4. Body mass index (BMI) of 18.5 to 35 kg/m2 at screening (both values inclusive).
5. Stable weight, with no more than 5 kg gain or loss in the 3 months prior to screening, this information will be collected by subject interview during medical history.
6. Glycosylated hemoglobin (HbA1c) ≤ 9.5% at screening.
7. Hemoglobin ≥9.0 g/dL at screening.
8. Subject has the capability of communicating appropriately with the investigator.
9. Subject is able and willing to comply with the requirements of the study protocol including the 8-point self-monitored blood glucose (SMBG), completion of subject diary records and following a recommended diet and exercise plan for the entire duration of the study.
10. Female subjects of childbearing potential who are willing to use oral contraception or two acceptable methods of contraception, (e.g., intra-uterine device plus condom, spermicidal gel plus condom, diaphragm plus condom, etc.), from the time of screening and for the duration of the study, through study completion.

    1. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    2. Postmenopausal females must have had no regular menstrual bleeding for at least 1 year prior to screening.
    3. Female subjects who report surgical sterilization must have had the procedure at least 6 months prior to screening.
    4. All female subjects of childbearing potential must have negative pregnancy test results at screening and at clinic visits, as per the SCHEDULE OF ACTIVITIES (SOA).
    5. If female subjects have male partners who have undergone vasectomy, the vasectomy must have occurred more than 6 months prior to screening

Exclusion Criteria:

1. History or presence of a medical condition or disease that in the investigator's opinion would place the subject at an unacceptable risk from study participation.
2. History of hypersensitivity to any of the active or inactive ingredients of the insulin/insulin analogue preparations used in the study, OR history of significant allergic drug reactions.
3. History of use of animal insulin within the last 3 years or use of approved biosimilar insulin glargine at any time prior to study entry, except for subject who previously participated in MYL-1501D studies and were compliant with the study protocols.
4. History of use of a regular immunomodulator therapy in the 1 year prior to screening.
5. History of autoimmune disorders other than T1DM or insufficiently treated autoimmune thyroid disorders judged clinically relevant by the investigator (recorded while collecting subject history).
6. History of ≥1 episodes of diabetic ketoacidosis or emergency room visits for uncontrolled diabetes leading to hospitalization within the 6 months prior to screening.
7. History of clinically significant acute bacterial, viral or fungal systemic infections in the last 4 weeks prior to screening (recorded while collecting subject history).
8. Any clinically significant abnormality in electrocardiogram (ECG) or safety laboratory tests (LFT, RFT, hematology or any other laboratory deemed clinically relevant by the investigator) conducted at screening and considered by the investigator to make the subject ineligible for the study.
9. Serological evidence of human immunodeficiency virus (HIV), hepatitis B surface antigen (HbSAg) or hepatitis C antibodies (HCVAb) at screening.
10. History of drug or alcohol dependence or abuse during the 1 year prior to screening.
11. Receipt of another investigational drug in the 3 months prior to screening (or as per local regulations), or if the screening visit is within 5 half-lives of another investigational drug received (whichever is longer), or scheduled to receive another investigational drug during the current study period.
12. Subjects with the following secondary complications of diabetes:

    1. Active proliferative retinopathy as confirmed by a dilated ophthalmoscopy examination / retinal photography (performed by a person legally authorized to do so) within the 6 months prior to screening.
    2. Clinical nephrotic syndrome or diabetic nephropathy with a serum creatinine level >1.5 times of upper limit of reference range at screening
    3. History of severe form of neuropathy or cardiac autonomic neuropathy, recorded while collecting subject history. Subject's with mild or moderate forms of neuropathy will be allowed.
    4. Subjects with a history of limb amputation as a complication of diabetes (at any time), or any vascular procedure during the 1 year prior to screening.
    5. History of diabetic foot or diabetic ulcers in the 1 year prior to screening.
13. Any elective surgery requiring hospitalization planned during the study period.
14. Clinically significant major organ disorder at the time of screening including:

    1. Uncontrolled hypertension, defined as stage 2 hypertension by Joint National Committee VII (even if therapy is ongoing, blood pressure ≥160 mm Hg systolic or ≥100 mm Hg diastolic).
    2. Uncontrolled hyperlipidemia (even if therapy is ongoing, LDL >160 mg/dL or triglycerides >500 mg/dL).
    3. Uncontrolled hyperthyroidism or hypothyroidism (subjects can be included if these conditions are controlled with thyroid hormones or anti-thyroid drugs).
    4. Impaired hepatic function (alanine transaminase [ALT] or aspartate transaminase [AST] value >2 times the upper limit of the reference range and/or serum bilirubin 1.5 times the upper limit of the reference range at the screening visit). Subjects with evidence of Gilberts disease may be included in the study if they have total bilirubin of <3 mg/dL with indirect bilirubin contributing to >80% of the total bilirubin.
15. History of a significant medical condition, such as:

    1. Clinically significant cardiac disease like unstable angina, myocardial infarction, grade 3 or 4 congestive heart failure (CHF) according to New York Heart Association criteria, valvular heart disease, cardiac arrhythmia requiring treatment, and pulmonary hypertension; during the year prior to screening.
    2. Stroke or transient ischemic attack (TIA) in the 6 months before screening.
16. Subjects with major depressive illness in the last 3 years (those who have well-controlled depression for 3 months on a stable dose of antidepressants, with no major depressive episodes in the last 3 years, can be included, even if they are on medication), subjects with history of other severe psychiatric diseases (manic depressive psychosis [MDP], schizophrenia), which in the opinion of the investigator precludes the subject from participating in the study (recorded while collecting subject history).
17. History of hematological disorders that can affect the reliability of HbA1c estimation (hemoglobinopathies, hemolytic anemia, sickle cell anemia, etc.).
18. Subjects using the following in the 3 months prior to screening:

    1. Insulin pump therapy
    2. Any anti-diabetic drugs other than the study insulins allowed by the protocol.
19. Moderate insulin resistance, defined as requiring insulin of ≥1.5 U/IU/kg/day.
20. Subjects who have received ≥14 consecutive days of glucocorticoid therapy by oral, intravenous, inhaled or other routes that produce systemic effects within the past 1 year, or who have received steroids by any route (except intra-nasal, intra-ocular, and topical) within the 4 weeks immediately preceding screening.
21. Subjects diagnosed as having cancer (subjects with history of basal cell carcinoma, carcinoma in situ or squamous cell cancer of skin, or in remission >5 years, will be allowed).
22. Subjects who have donated blood or plasma in the 1 month prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2019-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - Mylan Investigator Site, Fresno, California
  - Mylan Investigator Site, Greenbrae, California
  - Mylan Investigator Site, Huntington Beach, California
  - Mylan Investigator Site, La Mesa, California
  - Mylan Investigator Site, Los Gatos, California
  - Mylan Investigator Site, Mission Hills, California
  - Mylan Investigator Site, Montclair, California
  - Mylan Investigator Site, Northridge, California
  - Mylan Investigator Site, Oakland, California
  - Mylan Investigator Site, Santa Monica, California
  - Mylan Investigator Site, Tarzana, California
  - Mylan Investigator Site, Tustin, California
  - Mylan Investigator Site, Walnut Creek, California
  - Mylan Investigator Site, Denver, Colorado
  - Mylan Investigator Site, Bradenton, Florida
  - Mylan Investigator Site, Fort Lauderdale, Florida
  - Mylan Investigator Site, Fort Myers, Florida
  - Mylan Investigator Site, Hialeah, Florida
  - Mylan Investigator Site, Maitland, Florida
  - Mylan Investigator Site, Miami, Florida
  - Mylan Investigator Site, New Port Richey, Florida
  - Mylan Investigator Site, Palm Harbor, Florida
  - Mylan Investigator Site, Spring Hill, Florida
  - Mylan Investigator Site, St. Petersburg, Florida
  - Mylan Investigator Site, Tampa, Florida
  - Mylan Investigator Site, West Palm Beach, Florida
  - Mylan Investigator Site, Atlanta, Georgia
  - Mylan Investigator Site, Columbus, Georgia
  - Mylan Investigator Site, Lawrenceville, Georgia
  - Mylan Investigator Site, Roswell, Georgia
  - Mylan Investigator Site, Idaho Falls, Idaho
  - Mylan Investigator Site, Meridian, Idaho
  - Mylan Investigator Site, Springfield, Illinois
  - Mylan Investigator Site, Council Bluffs, Iowa
  - Mylan Investigator Site, Austin, Texas
  - Mylan Investigator Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MYL-1501D (Process V Product): MYL-1501D (Process V Product)
  MYL-1501D: Process V or Process VI
- MYL-1501D (Process VI Product): MYL-1501D (Process VI Product)
  MYL-1501D: Process V or Process VI
Period: Overall Study
Arm/Group | MYL-1501D (Process V Product) | MYL-1501D (Process VI Product)
Started | 108 | 111
Completed | 103 | 102
Not Completed | 5 | 9
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Per sponsor due to noncompliance | 1 | 0
Not completed — Subject off study medication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MYL-1501D (Process V Product) | MYL-1501D (Process VI Product) | Total
Number analyzed (Participants) | 108 | 111 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (11.46) | 42.8 (12.14) | 42.8 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 71
  Male | 72 | 76 | 148
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 11 | 18
  Not Hispanic or Latino | 98 | 98 | 196
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 95 | 103 | 198
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Screening Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 83.58 (16.137) | 82.42 (14.782) | 82.99 (15.441)
Screening BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 27.37 (3.726) | 27.29 (3.927) | 27.33 (3.821)
Duration of diabetes [Mean (Standard Deviation); unit: years] | 22.321 (13.2876) | 21.736 (13.3418) | 22.025 (13.2878)
Time of glargine administration [Count of Participants; unit: Participants]
  Morning | 32 | 37 | 69
  Evening | 76 | 74 | 150
Baseline FPG [Mean (Standard Deviation); unit: mmol/L] | 8.793 (3.9095) | 9.065 (3.7223) | 8.931 (3.8094)
Baseline HbA1c [Mean (Standard Deviation); unit: %] | 7.281 (0.8759) | 7.371 (0.8681) | 7.327 (0.8711)
Insulin use prior to screening [Count of Participants; unit: Participants]
  Yes | 108 | 111 | 219
  No | 0 | 0 | 0
Fasting C-peptide [Mean (Standard Deviation); unit: mmol/L] | 0.041 (0.0430) | 0.039 (0.0533) | 0.040 (0.0484)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Change in HbA1c from baseline
Time Frame: Baseline to Week 18
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | MYL-1501D (Process V Product) | MYL-1501D (Process VI Product)
Number analyzed (Participants) | 108 | 111
percentage of change | 0.18 (0.055) | 0.15 (0.053)

2. Secondary Outcome: Change in FPG
Description: Change in fasting plasma glucose from baseline
Time Frame: Baseline to Week 18
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MYL-1501D (Process V Product) | MYL-1501D (Process VI Product)
Number analyzed (Participants) | 108 | 111
mmol/L | 0.64 (5.754) | 0.01 (4.767)

3. Secondary Outcome: Change in Insulin Dose
Description: Change in daily total insulin dose per unit body weight (U/kg) from baseline
Time Frame: Baseline to Week 18
Measure: Mean (Standard Deviation); unit: Units per kilogram
Arm/Group | MYL-1501D (Process V Product) | MYL-1501D (Process VI Product)
Number analyzed (Participants) | 108 | 111
Units per kilogram | -0.004 (0.1039) | 0.007 (0.0884)

4. Secondary Outcome: Change in 8-point SMBG
Description: Change in 8-point self-monitored blood glucose (SMBG) daily average
Time Frame: Baseline to Week 18
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MYL-1501D (Process V Product) | MYL-1501D (Process VI Product)
Number analyzed (Participants) | 108 | 111
mmol/L | 0.10 (1.317) | 0.11 (1.743)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of signing Informed Consent through completion of the Follow-up visit, an average of 26 weeks. All safety analyses were carried out using the Safety population, which was defined as all subjects who were randomized and received ≥ 1 dose of IP.
Arm/Group | MYL-1501D (Process V Product) | MYL-1501D (Process VI Product)
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/110
Serious Adverse Events (participants affected / at risk) | 3/108 | 7/110
Other Adverse Events (participants affected / at risk) | 45/108 | 46/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MYL-1501D (Process V Product) (N=108) | MYL-1501D (Process VI Product) (N=110)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (4) | 4 (4)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MYL-1501D (Process V Product) (N=108) | MYL-1501D (Process VI Product) (N=110)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (5) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 3 (3)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4)
Gastroenteritis (Infections and infestations) | 4 (5) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (4) | 4 (4)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Left atrial enlargement (Cardiac disorders) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (5) | 5 (6)
Gastrooesophagael reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Genital herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Injection site infection (Infections and infestations) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pyuria (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Root canal infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Viral respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Weight increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 2 (2) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vasectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT03376789/Prot_001.pdf
  • Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT03376789/SAP_000.pdf